CLINICAL TRIAL: NCT01807039
Title: Mortality Following Surgery for Proximal Femoral Fractures
Acronym: HipMo
Status: Completed | Type: Observational
Sponsor: Brno University Hospital (Other)
Collaborators: St. Anne's University Hospital Brno, Czech Republic (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, MD, Ph.D., Brno University Hospital
Other Study IDs: KARIM FN Brno
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Fracture of Neck of Femur (Hip)
Keywords: hip fracture; proximal femur; pertrochanteric fracture; subtrochanteric fracture; subcapital fracture; safety issue; anesthesia
MeSH Terms: conditions — Femoral Neck Fractures; Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients after surgery with isolated proximal femur fracture: Patients between 18-110 years admitted to Faculty Hospital Brno with isolated injury of proximal femur (ICD dg. S72.0 a S72.1)who underwent surgery between 1.1. 2011 00:00 - 31.12. 2012 23:59 in Faculty hospital Brno (tertiary care university hospital).
  Interventions: Procedure: hip fracture surgery

INTERVENTIONS:
Procedure: hip fracture surgery — we evaluate the relationship between the monitored parameters and 30 day survival

SUMMARY:
Proximal femoral fractures are most frequent traumatologic and orthopedic diagnoses undergoing surgery. It affect most seniors and accompanied by a series of complications. The aim of our retrospective clinical trial is to establish a thirty-day mortality rate after surgical solutions, mortality during hospitalization and compare the types of anesthesia chosen during the performance (general vs. subarachnoid anesthesia).

DETAILED DESCRIPTION:
We evaluate relationship between the monitored parameters and 30 day survival.

Observed parameters:

* age of the patient
* sex of the patient
* 90 days mortality rate
* American Society of Anesthesiologists (ASA) score
* time since injury and surgery (hours)
* whether surgery was initiated during the day (7:00 - 20:00) or at night (20:00-07:00)
* type of administered anesthesia (GA, epidural anaesthesia, Subarachnoid (spinal) block)
* hemoglobin level prior to surgery
* haemotransfusion administration during surgery
* perioperative administration of vasopressors
* anesthetist erudition (with / without accomplished residency)
* surgeon erudition (with / without accomplished residency)

ELIGIBILITY:
Inclusion Criteria:

* isolated fracture of proximal femur indicated for surgery

Exclusion Criteria:

* children under 18 years
* none isolated trauma
* isolated fracture of proximal femur without surgery

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: isolated fracture of proximal femur indicated for surgery
Sampling Method: Probability Sample
Enrollment: 369 (Actual)
Dates: Start 2012-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
in hospital mortality rate | 2 years
  number of deaths from hospital admission to discharge (percent)

SECONDARY OUTCOMES:
30 days mortality rate | 2 years
  number of deaths within 30 days after injury (percent)

CONTACTS AND LOCATIONS:
Overall Officials: Petr Štourač, MD, Ph.D., Study Director — Brno Faculty Hospital, departement of anesthesiology and intensive care medicine
Locations (1):
- Faculty Hospital Brno, Brno, South Moravian, Czechia

REFERENCES:
- [Background] O'Hara DA, Duff A, Berlin JA, Poses RM, Lawrence VA, Huber EC, Noveck H, Strom BL, Carson JL. The effect of anesthetic technique on postoperative outcomes in hip fracture repair. Anesthesiology. 2000 Apr;92(4):947-57. doi: 10.1097/00000542-200004000-00011. PMID 10754613
- [Background] Pearse RM, Moreno RP, Bauer P, Pelosi P, Metnitz P, Spies C, Vallet B, Vincent JL, Hoeft A, Rhodes A; European Surgical Outcomes Study (EuSOS) group for the Trials groups of the European Society of Intensive Care Medicine and the European Society of Anaesthesiology. Mortality after surgery in Europe: a 7 day cohort study. Lancet. 2012 Sep 22;380(9847):1059-65. doi: 10.1016/S0140-6736(12)61148-9. PMID 22998715
- [Background] Dzupa V, Bartonicek J, Skala-Rosenbaum J, Prikazsky V. [Mortality in patients with proximal femoral fractures during the first year after the injury]. Acta Chir Orthop Traumatol Cech. 2002;69(1):39-44. Czech. PMID 11951568
- See also: open access link to full-text — http://www.achot.cz/detail.php?stat=769